CLINICAL TRIAL: NCT02323984
Title: Postoperative Delirium in Patients Undergoing Hip Arthroplasty
Brief Title: Postoperative Delirium in Hip Arthroplasty Patients
Acronym: mRNAOrtho
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Nicoleta Stoicea, Co-Principal Investigator, Ohio State University
Other Study IDs: 2013H0291
Record Dates: First submitted 2014-12-16; First posted 2014-12-24 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Delirium; Postoperative Complications
MeSH Terms: conditions — Delirium; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hypoactive Delirium - Delirious: Hypoactive delirious patients presenting with lethargy and sedation and are slow to respond to questions and demonstrate little spontaneous movement. miRNA Testing, Microemboli Monitoring, Delirium Assessment will be performed
  Interventions: Other: miRNA Testing, Microemboli Monitoring, Delirium Assessment
- Hyperactive Delirium - Delirious: Hyperactive delirious patients presenting with restlessness, agitation, hyper vigilance, and occaionally hallucinations. miRNA Testing, Microemboli Monitoring, Delirium Assessment will be performed
  Interventions: Other: miRNA Testing, Microemboli Monitoring, Delirium Assessment
- No Delirium - Nondelirious: Patients not presenting any symptoms of hypoactive or hyperactive postoperative delirium. miRNA Testing, Microemboli Monitoring, Delirium Assessment will be performed
  Interventions: Other: miRNA Testing, Microemboli Monitoring, Delirium Assessment

INTERVENTIONS:
Other: miRNA Testing, Microemboli Monitoring, Delirium Assessment — Delirium assessment questionnaire and blood testing for miRNA will be done for all patients postoperatively, as well as BIS monitoring during surgery. The three arms of the study indicate the allocation of each patient based on their delirium presentation (hypoactive, hyperactive, or none).

SUMMARY:
Identification of specific circulating microRNAs and microemboli formation (diagnosed by TC Doppler) in both delirious groups and nondelirious group will be our primary target. Delirium assessment through standardized questionnaires will be done at baseline (day of the surgery - pre operatory), immediately after surgery (in post anesthesia care unit) and then every 12 hours in Day 1 and Day2 after surgery. The investigators will use linear mixed models to describe the change patterns overtime, and compare differences at each time point. Inflammatory biomarkers will be explored overtime as well. The investigators will also explore age effect on cognitive function - cognitive reserve - based on the score of the cognitive test administered at baseline.

DETAILED DESCRIPTION:
Specific circulating microRNA's have been identified in patients with neurological diseases or deficits, and specifically those with neurodegenerative conditions. Furthermore, available evidence primarily in pre-clinical / animal models supports the hypothesis that post-surgical/anesthesia - induced neuroinflammation leads to post-operative cognitive decline or dysfunction. The investigators hypothesize that specific circulating microRNA's involved in the pro-inflammatory response to surgery/anesthesia are a suitable biomarker of Delirium and/or POCD in surgical hip-arthroplasty patients. However, it is also possible that microamboli during the surgical procedure could contribute to these neurologic outcomes. Therefore, in addition to analyzing microRNA levels (our primary target), the investigators propose to monitor cerebral vascular flow during the surgery to possibly identify microambolic events using Transcranial Doppler. Overall, our overarching goal is to identify novel early clinical indicators of cognitive dysfunction (e.g. Delirium and POCD).

The study will include preoperative-postoperative trajectory as well as the value of using subjects as self-controls with appropriate longitudinal analyses of cognition.

There are many factors that are potential confounders in relation to cognitive decline and incident dementia.

There are key characteristics and events:

* illnesses requiring hospitalization, that could potentially accelerate cognitive decline or worsen clinical dementia rating
* which anesthetic agents are administered for the surgical procedure
* intra-operative adverse events (anesthesia/surgery related, cerebral hypoxia, hypotension/hypertension, blood loss)
* patient factors (age, education, comorbidity)
* physiologic factors (inflammation,micro-embolization, blood-brain barrier function);
* perioperative factors (medications, sleep, complications)
* postoperative factors (rehabilitation, depression, social support)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 30 and 80 years of age
* ASA I , II or III
* Capable and willing to consent
* Participants literate in English language

Exclusion Criteria:

* ASA IV or V
* Patients with severe visual or auditory disorder
* Illiteracy
* Presence of a clinically diagnosed major psychiatric condition such as bipolar disorder, uncontrolled major depression, schizophrenia
* Dementia of Alzheimer's type
* Parkinson disease
* Multiple Sclerosis (MS)
* Vascular dementia

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects schedule to undergo hip arthroplasty surgery
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Identification of specific circulating microRNAs in post operative delirium patients | Baseline, perioperatively and during post operative hospitalization (Day 1 and Day 2 post surgery)
  Identification of specific circulating microRNAs and microemboli formation (diagnosed by TC Doppler) in both delirious groups and nondelirious group will be our primary target. Our overarching goal is to identify novel early clinical indicators of cognitive dysfunction (e.g. Delirium and POCD)

SECONDARY OUTCOMES:
Age effects on cognitive function (cognitive reserve) | Baseline
  We will explore age effect on cognitive function (cognitive reserve), based on the baselin cognitive assessment score.

CONTACTS AND LOCATIONS:
Overall Officials: Fievos L Christofi, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States